CLINICAL TRIAL: NCT06861400
Title: Self-Reflective Resilience-Recovery Activity Promotion Training for Emergency Medical Service Personnel
Brief Title: A Digital Resilience Intervention for Emergency Medical Service Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse University (Other)
Responsible Party: Principal Investigator, Bryce Hruska, Associate Professor, Syracuse University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 11-3278-2022
Record Dates: First submitted 2025-02-24; First posted 2025-03-06 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Feasibility; Acceptability; Adoptability; Meaning Made; Adaptive Self-reflection; Recovery Activities; Recovery Experiences; Post Traumatic Stress Disorder PTSD; Anxiety; Depression
Keywords: Emergency Medical Service Personnel; Psychological Resilience
MeSH Terms: conditions — Combat Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-Reflective Resilience-Recovery Activity Promotion Training (SRR-RAPT) (Experimental): Receives Self-Reflective Resilience-Recovery Activity Promotion Training (SRR-RAPT)
  Interventions: Behavioral: Self-Reflective Resilience-Recovery Activity Promotion Training
- Usual Care (No Intervention): Does not receive SRR-RAPT.

INTERVENTIONS:
Behavioral: Self-Reflective Resilience-Recovery Activity Promotion Training — Self-Reflective Resilience-Recovery Activity Promotion Training (SRR-RAPT) promotes finding positive meaning in stressors by building self-awareness of the coping and regulatory responses used to manage them; evaluating those responses; adapting them based upon their perceived effectiveness; and developing a plan for managing similar stressors in the future based on what can be learned from the current situation. In addition to prompting self-monitoring and active reflection on stressors and coping responses, SRR-RAPT encourages practicing recovery activities that permit a person's stressor induced strain level to return to baseline. SRR-RAPT is administered daily for 8 consecutive days.
  Arms: Self-Reflective Resilience-Recovery Activity Promotion Training (SRR-RAPT)

SUMMARY:
Emergency medical service (EMS) workers (i.e., ambulance service providers) experience triple the risk for anxiety, depression, and posttraumatic stress disorder (PTSD) compared to the general U.S. population. These mental disorders impact health and well-being across the life course. Thus, there is a critical need for interventions targeting key risk factors that can reduce EMS workers' mental health risk. Chronic stress represents such a risk factor and is a routine feature of the EMS profession due to the demands of providing emergency medical care. Self-Reflective Resilience-Recovery Activity Promotion Training (SRR-RAPT) promotes finding positive meaning in stressors by building self-awareness of the coping and regulatory responses used to manage them; evaluating those responses; adapting them based upon their perceived effectiveness; and developing a plan for managing similar stressors in the future based on what can be learned from the current situation. In addition to prompting self-monitoring and active reflection on stressors and coping responses, SRR-RAPT encourages practicing recovery activities that permit a person's stressor induced strain level to return to baseline. The primary objective of the current study is to evaluate the feasibility, acceptability, and adoptability of SRR-RAPT among EMS personnel. A secondary objective was to examine the intervention's effect on hypothesized mechanisms of action predicted to vary in response to the intervention, as well as consider the intervention's ability to reduce mental health symptoms. It is hypothesized that the intervention will be associated with more positive meaning made, adaptive self-reflection, recovery activities, and recovery experiences, as well as lower levels of mental health symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Full-time or part-time employee at an emergency medical service agency
* ≥ 18 years of age
* ≥ 1 emergency medical service shift scheduled in the next 8 days from recruitment date.

Exclusion Criteria:

* Not a full-time or part-time employee at an emergency medical service agency
* < 18 years of age
* < 1 emergency medical service shift scheduled in the next 8 days from recruitment date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Time period required to achieve target sample size | From study initiation until at least 80 participants are recruited, up to 12 months
  The number of months it takes to recruit the number of participants necessary to reach the target sample size.
Number of participants recruited and randomized each week of the study | From study initiation until at least 80 participants are recruited, up to 12 months
  A count of the number of participants who are recruited and randomized each week that the study is taking place.
Acceptability | Day 8 of the intervention
  Assessed with 3 items asking about respondents' perceptions that the intervention was helpful ("I found that answering the questions about managing stressful experiences and practicing recovery behaviors was helpful"); useful ("I found that answering the questions about managing stressful experiences and practicing recovery behaviors was useful"); and not burdensome ("I found that answering the questions about managing stressful experiences and practicing recovery behaviors was not too burdensome"). Respondents rated each item on a scale ranging from 1 ("Strongly Disagree") to 5 ("Strongly Agree"). Ratings are summed to yield a total daily score.
Adoptability | Day 8 of the intervention
  Assessed with 3 items asking about respondents intention to use what they had learned from the intervention in the future ("I will keep using these questions to help manage stressful experiences and practice recovery activities in the future." "I will try to use these questions in the future when managing stressful experiences and trying to practice recovery activities." "I plan to use some of the approaches that I came up with in my responses to the questions about managing stressful experiences and practicing recovery behaviors in the future"). Respondents rate each item on a scale ranging from 1 ("Strongly Disagree") to 5 ("Strongly Agree"). Ratings are summed to yield a total daily score.

SECONDARY OUTCOMES:
Meaning Made | Days 1 to 8 of the intervention
  Assessed using 3 items with the highest factor loadings on the positive reframing, acceptance, and religion subscales of the Brief COPE plus one additional item representing growth ("I identified lessons that I can learn from the challenge"). Respondents rate how much they performed the strategy described in response to any stressful or challenging experiences they encountered today. Ratings are made on a scale ranging from 1 ("Not at all") to 4 ("I did this a lot"). Ratings are summed to yield a total daily score.
Adaptive Self-Reflection | Days 1 to 8 of the intervention
  Derived from 3 items used in prior research. Each day respondents rate how much they agree with the following statements describing how they reacted to challenging and stressful events they encountered today: "I noticed the strategies that I used to cope with today's stress experiences", "I considered how I approach stressful experiences in my life", and "After attempting to deal with any of today's stressful experiences, I thought about how well my approach worked." Ratings are made on a scale ranging from 1 ("Strongly Disagree") to 5 ("Strongly Agree"). Ratings are summed to yield a total daily score.
Recovery Activities | Days 1 to 8 of the intervention
  Pittsburgh Enjoyable Activities Test. For each item, respondents indicate whether they did the activity described today when they were not working ("Yes" vs "No"). Endorsed items are summed to yield a total daily count.
Recovery Experiences | Days 1 to 8 of the intervention
  Derived from 8 items with the highest factor loadings from the detachment, relaxation, mastery, and control subscales of the Recovery Experiences Questionnaire. Respondents report how much they agree with each statement describing what they did during their off-job time today on a scale ranging from 1 ("Totally Disagree") to 5 ("Totally Agree"). Ratings are summed to yield a total daily score.
PTSD Symptom Severity | Days 1 to 8 of the intervention
  Short -form of the PTSD Checklist for DSM-5. Each day respondents rate how bothered they are by PTSD symptoms on a scale ranging from 0 ("Not at all") to 4 ("Extremely"). Ratings are summed to yield a total daily score.
Depression Symptom Severity | Days 1 to 8 of the intervention
  PROMIS-dep-4a questionnaire. Each day respondents rate the extent they experienced depression symptoms on a scale ranging from 1 ("Not at all") to 5 ("All of the time"). Ratings are summed to yield a total daily score.
Anxiety Symptom Severity | Days 1 to 8 of the intervention
  PROMIS-anx-4a questionnaire. Each day respondents rate the extent they experienced anxiety symptoms on a scale ranging from 1 ("Not at all") to 5 ("All of the time"). Ratings are summed to yield a total daily score.

CONTACTS AND LOCATIONS:
Locations (1):
- Syracuse University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cella D, Choi SW, Condon DM, Schalet B, Hays RD, Rothrock NE, Yount S, Cook KF, Gershon RC, Amtmann D, DeWalt DA, Pilkonis PA, Stone AA, Weinfurt K, Reeve BB. PROMIS(R) Adult Health Profiles: Efficient Short-Form Measures of Seven Health Domains. Value Health. 2019 May;22(5):537-544. doi: 10.1016/j.jval.2019.02.004. PMID 31104731
- [Background] Zuromski KL, Ustun B, Hwang I, Keane TM, Marx BP, Stein MB, Ursano RJ, Kessler RC. Developing an optimal short-form of the PTSD Checklist for DSM-5 (PCL-5). Depress Anxiety. 2019 Sep;36(9):790-800. doi: 10.1002/da.22942. Epub 2019 Jul 29. PMID 31356709
- [Background] Sonnentag S, Fritz C. The Recovery Experience Questionnaire: development and validation of a measure for assessing recuperation and unwinding from work. J Occup Health Psychol. 2007 Jul;12(3):204-21. doi: 10.1037/1076-8998.12.3.204. PMID 17638488
- [Background] Pressman SD, Matthews KA, Cohen S, Martire LM, Scheier M, Baum A, Schulz R. Association of enjoyable leisure activities with psychological and physical well-being. Psychosom Med. 2009 Sep;71(7):725-32. doi: 10.1097/PSY.0b013e3181ad7978. Epub 2009 Jul 10. PMID 19592515
- [Background] Cooper C, Katona C, Livingston G. Validity and reliability of the brief COPE in carers of people with dementia: the LASER-AD Study. J Nerv Ment Dis. 2008 Nov;196(11):838-43. doi: 10.1097/NMD.0b013e31818b504c. PMID 19008735
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744